CLINICAL TRIAL: NCT06736769
Title: "KETTLE" Trial: Ketamine Effects on Learning In Eating Disorders
Brief Title: Ketamine Effects on Learning In Eating Disorders
Acronym: KETTLE
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Amanda Downey, MD (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Amanda Downey, MD, Assistant Professor of Pediatrics and Psychiatry and Behavioral Sciences, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL2TR001870 (NIH); KL2TR001870 (NIH); P0541014 (Other: UCSF Clinical and Translational Science Institute (CTSI) Proposal Number); 24--42123 (Other: UCSF Institutional Review Board Number)
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Anorexia Nervosa; Atypical Anorexia Nervosa
Keywords: Anxiety; Depression; Anorexia; Psychotropic Drugs; Feeding and Eating Disorders; Physiological Effects of Drugs; Cognitive Flexibility
MeSH Terms: conditions — Anorexia Nervosa; Anxiety Disorders; Depression; Anorexia; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine Infusion (Experimental)
  Interventions: Drug: Ketamine infusion

INTERVENTIONS:
Drug: Ketamine infusion — Ketamine will be delivered intravenously at 0.5 mg/kg over 40 minutes.

SUMMARY:
This is a single site, single dose clinical trial of intravenous (IV) ketamine for medically hospitalized adolescents and young adults with anorexia nervosa or atypical anorexia nervosa. Eating disorder symptoms will be measured pre- and post-ketamine infusion. Investigators hypothesize that ketamine will increase cognitive flexibility, making medical hospitalizations less distressing by improving the ability to learn new, positive associations with food.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-26 years old
2. Meets diagnosis of anorexia nervosa (AN) or atypical anorexia nervosa (atypical AN) per DSM-5 criteria on admission
3. Admitted to the medical hospital for malnutrition
4. No changes to psychiatric medications for month prior to trial enrollment
5. Agree to use a highly effective form of contraception for at least two weeks following ketamine administration
6. Have an outpatient primary care provider, medical provider, or behavioral health provider or psychiatrist who is actively managing or coordinating care

Exclusion Criteria:

1. Lifetime history of any psychotic disorder
2. Moderate or severe substance use disorder
3. Pregnancy as indicated by a positive urine pregnancy test during screening, lactation, or the intention of becoming pregnant within 3 months of entry into this trial
4. Electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) treatment within 30 days prior to enrollment
5. Intellectual or developmental disability
6. High risk for self-harm/suicide
7. Active laxative misuse or abuse
8. Biochemical refeeding syndrome or electrolyte abnormality
9. Cardiac abnormalities identified on admission
10. Taking medications that would be unsafe to administer with ketamine
11. Other medical condition or diagnosis, physical exam finding, laboratory abnormality, or health risk that would increase the risk of adverse events, at the discretion of the investigators

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean Change From Baseline in Reversal Learning | Day 2, Day 4
  Mean change in reversal learning as measured by the probabilistic reversal learning task.In the task, participants are presented with two stimuli, told to choose one of the two stimuli on each trial, and receive feedback regarding whether the stimulus is "Correct" or "Incorrect." Participants must modify their choice based on c hanging stimulus-outcome contingencies over time, engaging flexible learning.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E. Downey, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No